CLINICAL TRIAL: NCT01285934
Title: A Trial of High Dose Immunosuppression and Autologous Hematopoietic Stem Cell Support Versus Intensive Insulin Therapy in Adults With Early Onset Type I Diabetes Mellitus
Brief Title: Hematopoietic Stem Cell Support Versus Insulin in T1D
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participant enrolled
Sponsor: Northwestern University (Other)
Collaborators: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diabetes2008
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hematopoietic Stem Cell Transplantation (Experimental): Patients who meet eligibility and have completed pre-HSCT testing in section 7.0 (study parameters) may be enrolled in the transplant arm and will undergo an Autologous Hematopoietic Stem Cell Transplantation
  Interventions: Biological: Autologous Hematopoietic Stem Cell Transplantation
- control arm of intensive insulin therapy (Other): The control arm of intensive insulin therapy (IIT) will enroll all patients who meet eligibility but decline HSCT or whose insurance does not approve payment for HSCT before expiration of eligibility (within 5 months of disease onset)
  Interventions: Drug: intensive insulin therapy

INTERVENTIONS:
Biological: Autologous Hematopoietic Stem Cell Transplantation — All participants randomized to the transplant arm wil undergo Autologous Hematopoietic Stem Cell Transplantation
  Arms: Hematopoietic Stem Cell Transplantation
Drug: intensive insulin therapy — The control arm will be either CSII via an insulin pump or intensive subcutaneous insulin therapy with multiple insulin injections (at least 4/day) utilizing a long acting background insulin and pre-meal rapid acting insulin.
  Other Names: IIT
  Arms: control arm of intensive insulin therapy

SUMMARY:
Type 1 diabetes mellitus (T1D) results from immune-mediated destruction of insulin-producing islet cells. The loss of islet cells is traditionally treated with insulin therapy and in some cases pancreas or islet cell transplantation. Another approach would be to preserve islet cell mass before it is irreversibly lost. Previous trials using immune suppression within 6 weeks of T1D onset have demonstrated diminished exogenous insulin requirements compared to untreated controls. In our prior phase I non-randomized study, by extending immune suppression to the point of immune ablation / immune reset with autologous HSC support, several patients with new onset T1D have maintained an insulin-free, drug free remissions for more than 4 years. Although these results appear highly promising, it may be argued that our results are mitigated by the documented honeymoon effect following T1D, that is by a normal transient insulin free interval occurring after disease onset in some patients. The goal of this trial is to extend this phase I study of new onset T1D to clarify whether our post transplant insulin free interval is due to treatment intervention (transplant) or a result of a normally occurring "insulin free honeymoon period". Both groups will receive identical change of life style (i.e. diet, exercise) education.

DETAILED DESCRIPTION:
Eligible patients will have type 1 diabetes (aged ≥ 18 years old) within five months of disease diagnosis, and a positive antibody to an islet cell autoantigen, and fasting C-peptide > 0.2 nmol/l. Hematopoietic stem cells will be mobilized with cyclophosphamide (2.0 g/m2) and granulocyte colony-stimulating factor (10 g/kg/day) collected from peripheral blood by leukoapheresis and cryopreserved. HSC will injected IV after conditioning with cyclophosphamide (200 mg/kg) divided 50 mg/kg on day -5, -4, -3, -2, and rabbit antithymocyte globulin (4.5 mg/kg) divided 0.5 mg/kg day-5, and 1.0 mg/kg day -4, -3-, -2, -1. Rituxan (500mg) IV will be given on days -6 and +1. The control arm will receive either continuous subcutaneous insulin infusion (CSII) or intensive subcutaneous insulin therapy with multiple insulin injections (at least 4/day) utilizing a long acting background insulin and pre-meal rapid acting insulin. The main outcome measure will be: fasting C-peptide. Other outcome measures will include: daily exogenous insulin requirements, serum levels of hemoglobin A1c, area under the curve (AUC) C-peptide levels during mixed meal tolerance test, islet cell autoantigen antibody titers, and quality of life (QOL) short form 36 (SF-36) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16 to 35 years old
* A diagnosis of type 1 diabetes by hyperglycemia and at least 1 antibody to islet cell autoantigen: GAD, IAA, ICA, IA-2, or Slc30A8
* Fasting C-peptide > 0.20 nmol / liter
* Enrollment within 5 months of T1D diagnosis
* Eligible patients must be referred to a fertility / reproductive endocrinologist and have written documentation of medical counseling advising patients about the risk of infertility and the possible options of sperm and oocyte banking before enrollment.

Exclusion Criteria:

* HIV positive
* Patients in the honeymoon phase not taking insulin
* Hepatitis A, B, or C positive
* On corticosteroids or other immune suppressive medications
* History of diabetic ketoacidosis
* Ongoing malignancy except localized treated basal cell or squamous skin cancer.
* History of cardiac disease or congestive heart failure or ventricular tachycardia or abnormal dobutamine cardiac echocardiogram
* Positive pregnancy test, inability or unwillingness to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a potential side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* DLCO < 60% of predicted
* Resting LVEF < 45%
* Creatinine > 1.5 mg/dl
* Known hypersensitivity to E Coli derived proteins.
* Transaminases greater than 2 times normal
* Positive tuberculosis skin test
* Any active infection
* Any co-morbid illness that in the opinion of the investigator would jeopardize the ability of the subject to tolerate the study.
* Failure to collect at least 2.0 x 106 CD34+ cells/kg
* History of alcohol or illicit drug abuse
* Unwilling to be compliant with change in life-style-diet and exercise

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
C-peptide | Every 6 months for 5 years
  C-peptide (fasting and every 30 minutes during 2 hour mixed meal tolerance test

SECONDARY OUTCOMES:
Insulin dose | 5 years
  Insulin dose, recorded as daily insulin dose in IU/Kg/day
Serum levels of hemoglobin A1c | 5 years
Stimulated C-peptide levels during mixed meal tolerance test | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University